CLINICAL TRIAL: NCT07118306
Title: A Multicenter Study of the Impact of a COPD Identification and Referral System on Patient Follow Up and Outcomes After an Acute COPD Exacerbation Resulting in an Emergency Department Visit or Hospitalization
Brief Title: COPD Exacerbation Follow Up
Status: Not yet recruiting | Type: Observational
Sponsor: Viz.ai, Inc. (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: VIZCOPD03
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Chronic obstructive pulmonary disease; Exacerbation; VizCOPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental Cohort: Prospective patients presenting to sites after implementation of the digital health tool.
- Control Cohort: Retrospective patients who presented to the same study sites under the standard of care clinical workflow before implementation of the digital health tool
- Exploratory Cohort: Patients who had no prior respiratory specialist follow up before implementation of the digital health tool and are re-assessed for follow up after implementation of the digital health tool.

SUMMARY:
The goal of this study is to evaluate the impact of implementing an AI-enabled clinical workflow tool (Viz COPD) on respiratory specialist follow up and clinical outcomes after an acute exacerbation.

DETAILED DESCRIPTION:
Time perspective: This study will collect data prospectively for the Experimental cohort and retrospectively for the Control cohort. There is also an Exploratory cohort which will collect retrospective and prospective data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older at the time of arrival to the emergency department.
* Patients with a clinical diagnosis of COPD who present to the emergency department for a moderate or severe COPD exacerbation.
* A moderate exacerbation is defined as an acute exacerbation requiring either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics.
* A severe exacerbation is defined as an acute exacerbation requiring hospitalization, or observation for >24 hours in emergency department/urgent care facility or resulting in death.
* Patients on dual (LABA/LAMA, LABA/ICS, LAMA/ICS) or triple (LABA/LAMA/ICS) long-acting bronchodilator inhalers.

Exclusion Criteria:

* Patients on bronchodilator inhaler monotherapy.
* Patients leaving against medical advice or expiring during hospitalization.
* Patients with tracheostomy.
* Patients with advanced cancer.
* Patients who have received a lung transplant.
* Discharge to hospice care.
* Transfer to another hospital.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target of five geographically dispersed U.S. hospital systems to capture a diverse patient population and COPD clinical workflow.
Sampling Method: Non-Probability Sample
Enrollment: 485 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of a digital health tool implementation on patient follow up with a respiratory specialist within 30 days after discharge for an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | From time of exacerbation to 30 days after discharge
  Proportion of patients with a respiratory specialist follow-up visit within 30 days after discharge in the experimental cohort compared to the control cohort.
To assess the effect of a digital health tool implementation on time to respiratory specialist follow-up after an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Up to 1 year
  Time from discharge to respiratory specialist follow-up visit in the experimental cohort compared to the control cohort.

SECONDARY OUTCOMES:
To assess the effect of a digital health tool implementation on patient follow up with a respiratory specialist within 90 days after discharge for an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment to 90 days after discharge
  Proportion of patients with a respiratory specialist follow-up visit within 90 days after discharge in the experimental cohort compared to the control cohort.
To assess the effect of a digital health tool implementation on readmission following an acute, severe COPD exacerbation. | Enrollment to 30 days after discharge
  Proportion of patients with all-cause readmission within 30 days after discharge in the experimental cohort compared to the control cohort.
To assess the effect of a digital health tool implementation on readmission following an acute, severe COPD exacerbation. | Enrollment to 90 days after discharge
  Proportion of patients with all-cause readmission within 90 days after discharge in the experimental cohort compared to the control cohort.
To compare exacerbation rate (moderate, moderate and severe, severe) in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment to 30 days after discharge
  Proportion of patients with an acute exacerbation (moderate, moderate and severe, severe) within 30 days after discharge in the experimental cohort compared to the control cohort
To compare exacerbation rate (moderate, moderate and severe, severe) in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment to 90 days post discharge
  Proportion of patients with an acute exacerbation (moderate, moderate and severe, severe) within 90 days after discharge in the experimental cohort compared to the control cohort
To compare exacerbation rate (moderate, moderate and severe, severe) in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment to 1 year post discharge
  Rate of acute exacerbations (moderate, moderate and severe, severe) at 1 year after discharge in the experimental cohort compared to the control cohort.
To compare healthcare resource utilization in the experimental and control cohort following discharge for an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment through 30 days after discharge
  Proportion of patients with a composite outcome consisting of emergency department visits, readmissions, or exacerbations within 30 days after discharge in the experimental cohort compared to the control cohort
To compare healthcare resource utilization in the experimental and control cohort following discharge for an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment through 90 days after discharge
  Proportion of patients with a composite outcome consisting of emergency department visits, readmissions, or exacerbations within 90 days after discharge inthe experimental cohort compared to the control cohort.
To compare healthcare resource utilization in the experimental and control cohort following discharge for an acute COPD exacerbation resulting in an emergency department visit or hospitalization - 1 year | Enrollment through 1 year after discharge
  Rate of a composite outcome consisting of emergency department visits, readmissions, or exacerbations at 1 year after discharge in the experimental cohort compared to the control cohort.
To compare the rate of cardiovascular events in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization - 30 days | Enrollment through 30 days after discharge
  Proportion of patients with a cardiovascular event within 30 days after discharge in the experimental cohort compared to the control cohort.
To compare the rate of cardiovascular events in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization - 1 year | Enrollment through 1 year after discharge
  Rate of cardiovascular events at 1 year after discharge in the experimental cohort compared to the control cohort.
To compare patient mortality in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization - 30 days | Enrollment through 30 days after discharge
  Proportion of patients with allcause mortality within 30 days after discharge in the experimental cohort compared to the control cohort
To compare patient mortality in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment through 90 days after discharge
  Proportion of patients with allcause mortality within 90 days after discharge in the experimental cohort compared to the control cohort.
To compare patient mortality in the experimental and control cohort after an acute COPD exacerbation resulting in an emergency department visit or hospitalization - 1 year. | Enrollment through 1 year after discharge
  Rate of all-cause mortality at 1 year after discharge in the experimental cohort compared to the control cohort.
To assess the impact of a digital health tool implementation on achieving pharmacological treatment that is consistent with the GOLD treatment recommendations after an acute COPD exacerbation resulting in an emergency department visit or hospitalization. | Enrollment through 90 days
  The proportion of patients in the experimental cohort with pharmacological treatment consistent with the GOLD treatment recommendations at 30 and 90 days after discharge for the index exacerbation compared to the control cohort.

IPD SHARING:
Plan to Share IPD: No